CLINICAL TRIAL: NCT05583916
Title: Phase I Safety and Feasibility Pilot Study of Same-Day Discharge After Video-Assisted Thoracoscopic Surgery (VATS) Anatomical Lung or Wedge Resection (VALUE Trial)
Brief Title: Same Day Discharge for Video-Assisted Thoracoscopic Surgery (VATS) Lung Surgery
Acronym: VALUE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Jonathan Spicer, Assistant Professor of Surgery, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-7318
Record Dates: First submitted 2022-10-04; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Lung Cancer; Surgery
Keywords: Same Day Discharge; Video-Assisted Thoracoscopic Surgery (VATS); Minimally Invasive Surgery; Enhanced Recovery Pathway
MeSH Terms: conditions — Lung Neoplasms | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung Cancer Patients (Other): Patients with stage I or II primary lung cancer or pulmonary metastasis scheduled to undergo surgery.
  Interventions: Procedure: Same Day Discharge - Video-Assisted Thoracoscopic Surgery (VATS) Lung

INTERVENTIONS:
Procedure: Same Day Discharge - Video-Assisted Thoracoscopic Surgery (VATS) Lung — All patients will be scheduled to surgery at the start of the day and will be discharged within the same day as the procedure.

SUMMARY:
Phase I to evaluate the safety and feasibility of same-day discharge in selected participants undergoing minimally-invasive lung surgery and who receive an enhanced recovery pathway.

ELIGIBILITY:
Inclusion Criteria:

* Signed or verbal informed consent by participant
* Male and female adults, age 18 and above
* Clinical stage I-II lung cancer (suspected, proven, unproven), or secondary pulmonary malignancy
* BMI < 35
* ECOG 0-1
* Eligible for surgery and lung cancer resection (FEV1 > 60%, DLCO > 60%)
* Elective VATS anatomic resection (segmentectomy or lobectomy), or wedge resection
* Capable caregiver for discharge home

Exclusion Criteria:

* Clinical stage III lung cancer
* Surgery requiring pneumonectomy
* Neoadjuvant therapy
* Active pregnancy or breastfeeding
* History of chronic pain syndromes
* History of chronic opioid use
* Concomitant major surgery indicated with current admission to hospital
* Anticipated intraoperative complication including conversion to thoracotomy, major bleeding requiring blood transfusion, extensive adhesiolysis, injury to mediastinal structures, airway injury, nerve injury (phrenic, recurrent)
* Need for epidural or patient-controlled intravenous analgesia
* Need for urinary catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Adverse Event Rate | 30 days post surgery
Same Day Discharge Rate | Throughout the trial, from start until completion of surgery for all the patients, up to 12 months.
Readmission Rate | 30 days post surgery
Rate of presentation to the emergency room after surgery | 30 days post surgery

SECONDARY OUTCOMES:
Edmonton Symptom Assessment Scale (ESAS) | 30 days post surgery
  Rating pain, fatigue, nausea, depression, anxiety, drowsiness, appetite, well-being and shortness of breath, on a scale of 1 to 10. Higher scores indicate more serious symptoms.
Functional Assessment of Cancer Therapy - Lung (FACT-L) | 30 days post surgery
  Rating questions regarding physical, social/family, emotion and function well-being as well as general questions regarding medical health, on a scale of 0-4 (from 'Not at all' to 'Very much').
Duration of indwelling chest tube catheter | 30 days post surgery or until the chest tube is removed (whichever comes last, assessed until 90 days post surgery)
Rate of screen failure | From trial start until last patient consented, up to 12 months.
  Feasibility calculation of the number of patients approached to participate compared to the number of patients consented to the trial.
Percent of eligible participants consented | From trial start until last patient consented, up to 12 months.
Pathway adherence rate | From moment of consent until 1 day post surgery.
  Calculation of the number of participants who stay on the same-day discharge pathway versus number of patients who deviate from the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Spicer, MD, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT05583916/Prot_000.pdf
  • Informed Consent Form (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT05583916/ICF_001.pdf